CLINICAL TRIAL: NCT00050687
Title: A Randomized, Serum Level-targeted Study Investigating the Safety and Pharmacokinetics of Orally Administered Gallium Maltolate in Patients With Various Refractory Malignancies
Brief Title: Safety and Pharmacokinetics of Orally Administered Gallium Maltolate in Various Refractory Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Titan Pharmaceuticals (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTP-370-01-01
Record Dates: First submitted 2002-12-17; First posted 2002-12-19 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2006-11

CONDITIONS: Prostatic Neoplasms; Multiple Myeloma; Bladder Neoplasms; Lymphoma
MeSH Terms: conditions — Prostatic Neoplasms; Multiple Myeloma; Urinary Bladder Neoplasms; Lymphoma | interventions — gallium maltolate

INTERVENTIONS:
Drug: Gallium maltolate

SUMMARY:
This study will test the safety, tolerance, and efficacy of different doses of oral gallium maltolate. Patients will receive oral gallium maltolate twice daily for 28-consecutive days followed by 14 days off treatment. This dosing cycle will be repeated. Adverse effects will be assessed and the levels of gallium in serum will be measured. Any effect of the drug on the cancer and any improvement in cancer-related symptoms will also be measured.

DETAILED DESCRIPTION:
Gallium maltolate is an orally bioavailable form of gallium. This is a safety, pharmacokinetic and preliminary efficacy study. The primary objective of the study is to assess the safety profile in patients after oral administration of different doses of gallium maltolate for up to six 42-day cycles (28 days of gallium maltolate, followed by 14 days off treatment). In addition, serum concentrations of gallium and associated pharmacokinetic variables will be measured. From this information, an optimal dose will be selected for assessment of anti-tumor efficacy. The study assesses the effects of oral administration of gallium maltolate on pain resulting from bony metastasis, on biochemical measures of bone turnover, and on disease progression and overall survival in patients with various refractory malignancies. Patients may receive up to 6 cycles of the investigational agent.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hormone refractory prostate cancer, refractory multiple myeloma, refractory bladder cancer, or malignant lymphoma;
* life expectancy of ≥6 months,
* Zubrod Performance Status of ≤2,
* adequate bone marrow function, renal function, liver function and pulmonary function;
* age ≥ 18 years;
* willing and able to give informed consent; and
* effective contraceptive use or non child-bearing potential.

Exclusion Criteria:

* 10% weight loss in the previous 3 months;
* active serious infection not controlled by antibiotics;
* initiation of bisphosphonates treatment within 30 days;
* participation in other research study within 30 days;
* uncontrolled brain metastasis,
* prior intrathecal chemotherapy or whole-brain radiotherapy,
* inability to comply with protocol or undergo specified tests;
* other active malignancy;
* optic neuritis, and
* routine use of diuretics (for initial phase of study only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-06; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Highlands Oncology Group, PA, Springdale, Arkansas
  - California Cancer Care, Greenbrae, California
  - Stanford University, Palo Alto, California
  - Southfield Oncology Institute, Southfield, Michigan
  - New York Presbyterian Hospital, New York, New York